CLINICAL TRIAL: NCT02989298
Title: Peritoneal Dialysis Registration System (PERSIST)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: PD registry
Record Dates: First submitted 2016-10-17; First posted 2016-12-12 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: ESRD; Disorders Associated With Peritoneal Dialysis
Keywords: Peritoneal Dialysis (PD); Residual renal function; Peritoneum function; Peritonitis rate; Technical survival; Patient survival
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The serum, urine, DNA and peritoneum tissue will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PD patients: End stage renal disease patients receiving peritoneal dialysis treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Registration of all PD patients in the First Affiliated Hospital of Sun Yat-sen University and other hospitals，which have signed the contract in China.

SUMMARY:
Brief Summary: The investigators are registering all PD patients at recruited hospitals and developing a PD database in China. Patients will be followed up every 3 months, and both baseline and follow-up information will be collected and input into the registration system. The patient survival, technical survival, peritonitis rate, longitudinal changes of residual renal function and peritoneum function, and quality of life for PD patients, etc, will be compared using the PD database.

DETAILED DESCRIPTION:
Detailed Description: The investigators are registering all end stage renal disease (ESRD) patients receiving peritoneal dialysis (PD) treatment, and developing a PD database in China. Patients' demographic characteristics (including age, gender, height, weight, BMI, smoking, drinking, and education, etc), clinical characteristics (primary cause of ESRD, dialysis prescription, patient's condition and lab measurements of serum, urine, and dialysate), drug information, complications and scores of quality of life at the baseline will be collected. Patients will be followed up every 3 months. Demographic and clinical characteristics, complications, drug information of patients will be collected at each visit. The patients' clinical outcomes, such as mortality (including all-cause mortality and cardiovascular disease mortality), technical survival, kidney transplantation, transfer to hemodialysis, hospitalization, occurrence of peritonitis, etc. were also followed up till the end of the study. The data of patient survival, technical survival, peritonitis rate, hospitalization rate, clinical lab parameters, longitudinal changes of residual renal function and peritoneum function, peritonitis rate, hospitalization rate, clinical lab parameters and quality of life for PD patients will be analyzed using the PD database.

ELIGIBILITY:
Inclusion Criteria:PD patients -

Exclusion Criteria:No

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients receiving PD treatment
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient survival of PD patients | 10 years
  Patient survival including all-cause and cardiovascular mortality.

SECONDARY OUTCOMES:
Technical survival of PD patients | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, M.D. & Ph.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China